CLINICAL TRIAL: NCT05293314
Title: Assessment of an Exhaled Breath Test Using High-Pressure Photon Ionization Time-of-Flight Mass Spectrometry to Detect Bronchiectasis
Brief Title: Assessment of an Exhaled Breath Test to Detect Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Chief of Respiratory and Critical Care Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20220303
Record Dates: First submitted 2022-03-14; First posted 2022-03-24 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-09

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; breathomics; exhaled breath
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — organic components in exhaled breath
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult patients with bronchiectasis (BE): Diagnosis of bronchiectasis was performed using chest HRCT scans in suspected patients with coughing and expectoration, or long durations of haemoptysis. High-resolution images were obtained during full inspiration at 1-mm collimation and 10-mm intervals from the apex to the base of the lungs. The presence of bronchiectasis was confirmed based on the following criteria: 1) lack of tapering in the bronchi; 2) dilation of the bronchi where the internal diameter was larger than that of the adjacent pulmonary artery; or 3) visualisation of the peripheral bronchi within 1 cm of the costal pleural surface or the adjacent mediastinal pleural surface.
  Interventions: Diagnostic Test: An exhaled breath test
- Healthy control group (HC): Control group is healthy participants.
  Interventions: Diagnostic Test: An exhaled breath test
- Unhealthy control group (UHC): Patients with interstitial lung disease or patients with Sarcoidosis. Interstitial lung disease is a heterogeneous pulmonary disease characterized with lung fibrosis and manifest with breathlessness. Sarcoidosis is a systemic disease of unknown etiology characterized by the formation of granulomas in various organs, mostly involved is the lungs and intrathoracic lymph nodes .
  Interventions: Diagnostic Test: An exhaled breath test

INTERVENTIONS:
Diagnostic Test: An exhaled breath test — All exhaled breath samples were collected by trained investigators following the same protocol. All participants fasted for at least 6 hours before breath collection. To reduce potential confounding factors, all participants were asked to not ingest spicy food, alcohol, or coffee the night before exhaled breath collection. Exhaled breath was collected in Tedlar air bags (DuPont de Nemours). The night before breath collection, the Tedlar bags were baked at 60 °C for 3 hours to fully release possible contaminants and continuously purged with high-purity nitrogen 4 times. Participants first gargled with pure water and then performed a single deep nasal inhalation followed by complete exhalation via their mouth into Tedlar bags. A total of 1000 mL of exhaled breath was collected from each participant. Breath sample detection was based on the HPPI-TOFMS platform.

SUMMARY:
To investigate whether the breath test is able to detect bronchiectasis using breathomics. This study was conducted with a prospective specimen collection, evaluator-blinded, case-controlled clinical study designed to evaluate the accuracy of breathomics to diagnosis of bronchiectasis in adults.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic airway inflammation with irreversible expansion of bronchial walls, which is characteristic by chronic cough, mucinous sputum, dyspnea and wheezing. High resolution CT (HRCT) combined with clinical manifestations is the main diagnostic method of bronchiectasis, but HRCT is expensive and radioactive. Therefore, it is urgent to develop a new technology to diagnose bronchiectasis. Exhaled breath may be a better tool for bronchiectasis detection because of its noninvasive nature. Many efforts have been made to develop breath tests for lung cancer, asthma and Helicobacter pylori infection. However, little studies pay attention to bronchiectasis. High-pressure photon ionization time-of-flight mass spectrometry (HPPI-TOFMS) is a promising tool for breath testing, because it is highly sensitive, does not require pretreatment of exhaled breath, and holds great tolerance for humidity. In our case-control diagnostic study, we investigated whether a breath test combining HPPI-TOFMS and a support vector machine (SVM) algorithm was able to distinguish patients with bronchiectasis from control individuals.

ELIGIBILITY:
Inclusion Criteria:

BE Patients were recruited according to the following inclusion criteria: (1) Age>18 years; (2) the diagnosis of BE was according to European Respiratory Society guidelines for the management of adult bronchiectasis; (3) Willing to join in and sign the informed consent form.

Healthy control subjects were recruited according to the following inclusion criteria:(1) Age>18 years; (2) No history of any lung disease (according to pulmonary imaging and physical examinations); (3) Willing to join in and sign the informed consent form.

Unhealthy control subjects were recruited according to the following inclusion criteria: (1) Age>18 years; (2) The diagnosis of ILD was according to HRCT and clinical symptoms by two experts' consensus; (3) The diagnosis of Sarcoidosis (SA) was according to American Thoracic Society Clinical Practice Guideline;(4) Willing to join in and sign the informed consent form.

Exclusion Criteria:

(1) Patients combined with serious comorbidities (chronic renal failure, hepatic disease, etc.); (2) Patients who are diagnosed with asthma, pneumonia, malignant tumor, and COPD; (3) Women who are pregnant or preparing for pregnancy or breastfeeding; (4) Participated in other clinical trials within three months; (5) Refused to join in and sign the informed consent form.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The age of all subjects were all older than 18 . The study population was recruited from Shanghai pulmonary hospital. Diagnosis of bronchiectasis was performed using chest HRCT scans in suspected patients with coughing and expectoration, or long durations of haemoptysis. Idiopathic bronchiectasis patients with acute exacerbation were included in the study. Healthy participants (HC) and unhealthy participants(UHC) were as control.
Sampling Method: Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, MD, Study Director — Department of Respiratory and Critical Care
Locations (1):
- Shanghai pulmonary hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Bronchiectasis: Diagnosis of bronchiectasis was performed using chest HRCT scans in suspected patients with coughing and expectoration, or long durations of haemoptysis. High-resolution images were obtained during full inspiration at 1-mm collimation and 10-mm intervals from the apex to the base of the lungs. The presence of bronchiectasis was confirmed based on the following criteria: 1) lack of tapering in the bronchi; 2) dilation of the bronchi where the internal diameter was larger than that of the adjacent pulmonary artery; or 3) visualisation of the peripheral bronchi within 1 cm of the costal pleural surface or the adjacent mediastinal pleural surface.
  an exhaled breath test: All exhaled breath samples were collected by trained investigators following the same protocol. All participants fasted for at least 6 hours before breath collection. To reduce potential confounding factors, all participants were asked to not ingest spicy food, alcohol, or coffee the night before exhaled breath collection. Exhaled breath was collected in Tedlar air bags (DuPont de Nemours). The night before breath collection, the Tedlar bags were baked at 60 °C for 3 hours to fully release possible contaminants and continuously purged with high-purity nitrogen 4 times. Participants first gargled with pure water and then performed a single deep nasal inhalation followed by complete exhalation via their mouth into Tedlar bags. A total of 1000 mL of exhaled breath was collected from each participant.
- Healthy Control Group: Control group is healthy participants.
  an exhaled breath test: All exhaled breath samples were collected by trained investigators following the same protocol. All participants fasted for at least 6 hours before breath collection. To reduce potential confounding factors, all participants were asked to not ingest spicy food, alcohol, or coffee the night before exhaled breath collection. Exhaled breath was collected in Tedlar air bags (DuPont de Nemours). The night before breath collection, the Tedlar bags were baked at 60 °C for 3 hours to fully release possible contaminants and continuously purged with high-purity nitrogen 4 times. Participants first gargled with pure water and then performed a single deep nasal inhalation followed by complete exhalation via their mouth into Tedlar bags. A total of 1000 mL of exhaled breath was collected from each participant.
- Unhealthy Control Group: Patients with interstitial lung disease or patients with Sarcoidosis. Interstitial lung disease is a heterogeneous pulmonary disease characterized with lung fibrosis and manifest with breathlessness. Sarcoidosis is a systemic disease of unknown etiology characterized by the formation of granulomas in various organs, mostly involved is the lungs and intrathoracic lymph nodes .
  an exhaled breath test: All exhaled breath samples were collected by trained investigators following the same protocol. All participants fasted for at least 6 hours before breath collection. To reduce potential confounding factors, all participants were asked to not ingest spicy food, alcohol, or coffee the night before exhaled breath collection. Exhaled breath was collected in Tedlar air bags (DuPont de Nemours). The night before breath collection, the Tedlar bags were baked at 60 °C for 3 hours to fully release possible contaminants and continuously purged with high-purity nitrogen 4 times. Participants first gargled with pure water and then performed a single deep nasal inhalation followed by complete exhalation via their mouth into Tedlar bags. A total of 1000 mL of exhaled breath was collected from each participant.
Period: Overall Study
Arm/Group | Patients With Bronchiectasis | Healthy Control Group | Unhealthy Control Group
Started | 228 | 231 | 85
Completed | 215 | 221 | 74
Not Completed | 13 | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Bronchiectasis | Healthy Control Group | Unhealthy Control Group | Total
Number analyzed (Participants) | 215 | 221 | 74 | 510
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [49 to 66] | 52 [46 to 59] | 65 [56 to 69] | 56 [48 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 145 | 33 | 328
  Male | 65 | 76 | 41 | 182
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI(Body Mass Index) [Median (Inter-Quartile Range); unit: kg/m^2] | 21.1 [19.1 to 23.2] | 23.9 [22 to 25.8] | 24.2 [22.5 to 26.7] | 22.9 [20.6 to 25.4]
Smoking [Count of Participants; unit: Participants]
  Smoker | 27 | 40 | 28 | 95
  Non-smoker | 183 | 162 | 46 | 391
  No record | 5 | 19 | 0 | 24
Alcohol [Count of Participants; unit: Participants]
  Drinker | 6 | 11 | 3 | 20
  Non-drinker | 204 | 173 | 71 | 448
  No record | 5 | 37 | 0 | 42

OUTCOME MEASURES:

1. Primary Outcome: The Ability of the Breath Test Model to Distinguish Bronchiectasis From Healthy People
Description: Evaluate the ability of the breath test model to distinguish bronchiectasis from healthy individuals by measuring the area under the receiver operating characteristic (ROC) curves. The maximum value in the area below the receiver is 1. The closer the value is to 1, the higher the prediction accuracy of the model.
Time Frame: One week.Exhaled breath samples were collected on the first day of patients' hospitalization and sent to detect VOCs.The entire process will take one week.
Population: All participants were randomly divided to a discovery cohort (n=252), an internal validation cohort (n=103) and a blinded test cohort (n=155). The main outcomes were assumed by the data analysed from the blinded test cohort which was mentioned above.
Measure: Count of Participants; unit: Participants
Groups:
- Bronchiectasis Participants: (1) Age>18 years, the diagnosis of bronchiectasis need reference to the definition of "idiopathic bronchiectasis" according to British Thoracic Society in 2010 or 2012 China bronchiectasis expert consensus; (2) Patients are clinically diagnosed as acute attack (AE) and need hospitalization, that is, they have the following three or more clinical symptoms within 48 hours: Cough; Changes in the amount or character of sputum; Purulent sputum; Shortness of breath or decreased exercise tolerance; weakness hemoptysis; (3) Patient quit smoking for more than two years; (4) Willing to join in and sign the informed consent form.
- Healthy Controls: (1) Age>18 years; (2) No history of any lung disease (except for the history of pneumonia in the past time and small pulmonary nodules); (3) Willing to join in and sign the informed consent form.
- Unhealthy Controls: Participants with interstitial lung disease or patients with Sarcoidosis.
Arm/Group | Bronchiectasis Participants | Healthy Controls | Unhealthy Controls
Number analyzed (Participants) | 215 | 221 | 74
Participants | 65 | 67 | 23
Statistical Analysis 1: Comparison: Bronchiectasis Participants vs Healthy Controls; Evaluate the ability of the breath test model to distinguish bronchiectasis from healthy individuals by measuring the area under the receiver operating characteristic (ROC) curves. The maximum value in the area below the receiver is 1. The closer the value is to 1, the higher the prediction accuracy of the model; Test type: Other — Evaluate the ability of the breath test model to distinguish bronchiectasis from healthy individuals by measuring the area under the receiver operating characteristic (ROC) curves. The maximum value in the area below the receiver is 1. The closer the value is to 1, the higher the prediction accuracy of the model; p < 0.05, Wilcoxon (Mann-Whitney); receiver operating characteristic = 0.964, 95% CI 2-sided [0.932 to 0.996]
Statistical Analysis 2: Comparison: Bronchiectasis Participants vs Unhealthy Controls; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Wilcoxon (Mann-Whitney); receiver operating characteristic = 0.932, 95% CI 2-sided [0.879 to 0.982]

2. Secondary Outcome: The Sensitivity of the Breath Test Model to Distinguish Bronchiectasis From Healthy People
Description: Sensitivity=number of true positives/(number of true positives+number of false negatives) * 100% Sensitivity is the rate of correctly judging patients.We calculated the sensitivity of the breath test model to distinguish bronchiectasis from healthy people.The maximum percentage of the sensitivity is 100%. The higher the percentage is , the more sensitive of the model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bronchiectasis Participants | Healthy Controls | Unhealthy Controls
Number analyzed (Participants) | 215 | 221 | 74
Participants | 65 | 67 | 23
Statistical Analysis 1: Comparison: Bronchiectasis Participants vs Healthy Controls; Sensitivity=number of true positives/(number of true positives+number of false negatives) * 100% Sensitivity is the rate of correctly judging patients.We calculated the sensitivity of the breath test model to distinguish bronchiectasis from healthy people.The maximum percentage of the sensitivity is 100%. The higher the percentage is , the more sensitive of the model; Test type: Other — Sensitivity=number of true positives/(number of true positives+number of false negatives) * 100% Sensitivity is the rate of correctly judging patients.We calculated the sensitivity of the breath test model to distinguish bronchiectasis from healthy people.The maximum percentage of the sensitivity is 100%. The higher the percentage is , the more sensitive of the model; Sensitivity = 86.2, 95% CI 2-sided [77.1 to 95.2]
Statistical Analysis 2: Comparison: Bronchiectasis Participants vs Unhealthy Controls; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; Sensitivity = 86.2, 95% CI 2-sided [77.1 to 95.2]

3. Other Pre Specified Outcome: The Specificity of the Breath Test Model to Distinguish Bronchiectasis From Healthy People
Description: Specificity=number of true negative cases/(number of true negative cases+number of false positive cases) * 100% The specificity is the rate of correctly judging non patients.We calculated the specificity of the breath test model to distinguish bronchiectasis from healthy people.The maximum percentage of the specificity is 100%. The higher the percentage is , the more specificity of the model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bronchiectasis Participants | Healthy Controls | Unhealthy Controls
Number analyzed (Participants) | 215 | 221 | 74
Participants | 65 | 67 | 23
Statistical Analysis 1: Comparison: Bronchiectasis Participants vs Healthy Controls; Specificity=number of true negative cases/(number of true negative cases+number of false positive cases) * 100% The specificity is the rate of correctly judging non patients.We calculated the specificity of the breath test model to distinguish bronchiectasis from healthy people.The maximum percentage of the specificity is 100%. The higher the percentage is , the more specificity of the model; Test type: Other — Specificity=number of true negative cases/(number of true negative cases+number of false positive cases) * 100% The specificity is the rate of correctly judging non patients.We calculated the specificity of the breath test model to distinguish bronchiectasis from healthy people.The maximum percentage of the specificity is 100%. The higher the percentage is , the more specificity of the model; Specificity = 92.5, 95% CI 2-sided [86.2 to 98.8]
Statistical Analysis 2: Comparison: Bronchiectasis Participants vs Unhealthy Controls; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; Specificity = 73.9, 95% CI 2-sided [56 to 91.9]

ADVERSE EVENTS:
Time Frame: 1 day
Description: If a participant experiences a progressive decrease in blood pressure or cardiac arrest within one day after being collected breath sample, we define a serious adverse event as occurring.
Arm/Group | Patients With Bronchiectasis | Healthy Control Group | Unhealthy Control Group
All-Cause Mortality (participants affected / at risk) | 0/215 | 0/221 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/215 | 0/221 | 0/74
Other Adverse Events (participants affected / at risk) | 5/215 | 0/221 | 2/74
OTHER ADVERSE EVENTS (reported when occurring in more than 0.196% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Bronchiectasis (N=215) | Healthy Control Group (N=221) | Unhealthy Control Group (N=74)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 — Only 2 of bronchiectasis participants and 1 of unhealthy controls cough transiently. However, they all returned to normal after taking a 10 minute break.
short of breath (Respiratory, thoracic and mediastinal disorders) | 3 | NA | 1 — Only 3 of bronchiectasis participants and 1 of unhealthy controls feel short of breath transiently. However, they all returned to normal after taking a 10 minute break.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT05293314/Prot_SAP_000.pdf